CLINICAL TRIAL: NCT03564795
Title: Effectiveness of KeraStat Gel for Improved Cosmesis of Partial Thickness Burns
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment
Sponsor: KeraNetics, LLC (Industry)
Collaborators: Wake Forest University (Other); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KSGL-CRD-003
Record Dates: First submitted 2018-06-11; First posted 2018-06-21 (Actual); Results first posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Partial-thickness Burn
Keywords: Wound Dressing; Keratin; Hydrogel; Burn Dressing

STUDY DESIGN:
Intervention Model Description: Randomized, controlled within-subject trial of 30 patients, each of whom will have a minimum of one burn treated with the KeraStat Gel device and one burn treated with the standard of care dressing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- KeraStat Gel (Experimental): Each enrolled subject will have at least one eligible burn randomized to the KeraStat Gel arm. This burn will be dressed with KeraStat Gel and covered by a secondary dressing. Subjects will be instructed to change the dressing and re-apply the KeraStat Gel per the instructions for use (at least every 3 days).
  Interventions: Device: KeraStat Gel
- Silver Sulfadiazine (Active Comparator): Each enrolled subject will have at least one eligible burn randomized to the Silver Sulfadiazine arm. This burn will be dressed with the Silver Sulfadiazine and covered by a secondary dressing. Subjects will be instructed to change the dressing and re-apply the Silver Sulfadiazine per the institution's Standard of Care instructions.
  Interventions: Device: Silver Sulfadiazine

INTERVENTIONS:
Device: KeraStat Gel — Wound dressing for partial thickness burns
  Arms: KeraStat Gel
Device: Silver Sulfadiazine — Wound dressing for partial thickness burns
  Other Names: SSD
  Arms: Silver Sulfadiazine

SUMMARY:
A randomized, controlled, 30-subject, within-subject trial for examining the effectiveness of KeraStat Gel, as opposed to the institutional standard of care, silver sulfadiazine, in improving cosmesis of the healed wound.

DETAILED DESCRIPTION:
The study seeks to determine whether the use of KeraStat Gel as the primary dressing for partial thickness burns results in improved cosmesis of the healed wound, and results in less painful dressing changes, faster reepithelialization, and reduction in need for excision and grafting. The study will enroll 30 subjects. The study design is a randomized, controlled, within-subject trial to compare the effectiveness of KeraStat Gel vs. standard of care (SOC), silver sulfadiazine (SSD). Each of two distinct burns will be randomized to the use of KeraStat Gel or SOC. Patients will be seen weekly for the first month and then at months 3, 6, and 12 post burn.

ELIGIBILITY:
Inclusion Criteria:

* Presenting with at least two comparable, discrete, and separate partial thickness thermal burns, as determined by the Investigator, measuring 50 - 1,000 cm2 each
* Study wounds identified are partial thickness depth
* KeraStat Gel and SSD can be applied to randomized study burn wounds as definitive care treatment within 24 hours from time of injury]
* Overall total body surface area burned < 20%

Exclusion Criteria:

* Pregnant or nursing
* Prisoner
* Presence of inhalation injury, as determined by the Investigator
* Injury requiring formal intravenous fluid resuscitation
* Concomitant non-thermal traumatic injuries
* Chronic medical conditions including, but not limited to, documented renal impairment (Cr > 2.5 mg/dL), hepatic impairment (Total bilirubin > 2.5 mg/dL), thromboembolic disorders, active infection in study wound areas, uncontrolled diabetes (HbA1C > 7%), HIV infection, history of melanoma or systemic malignancy within the last 10 years
* Receiving corticosteroids, immunosuppressive agents, radiation or chemotherapy, topical growth factors, or any other medication the Investigator feels will affect wound healing
* Not expected to live at least 13 months post-burn
* Received an investigational drug or biologic within 3 months prior to injury
* Previously treated with a skin graft at either of the treatment sites
* Chemical or electrical burn
* Known or documented allergy to sulfonamides
* Proposed study wounds are full thickness
* Any condition the Investigator determines will compromise subject safety or prevent the subject from completing the study

Ages: 6 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-08-31 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James H Holmes IV, MD, Principal Investigator — Wake Forest Burn Center
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wasiak J, Cleland H, Campbell F. Dressings for superficial and partial thickness burns. Cochrane Database Syst Rev. 2008 Oct 8;(4):CD002106. doi: 10.1002/14651858.CD002106.pub3. PMID 18843629
- [Background] Tandara AA, Mustoe TA. The role of the epidermis in the control of scarring: evidence for mechanism of action for silicone gel. J Plast Reconstr Aesthet Surg. 2008 Oct;61(10):1219-25. doi: 10.1016/j.bjps.2008.03.022. Epub 2008 Jul 23. PMID 18653391
- [Background] Mustoe TA, Gurjala A. The role of the epidermis and the mechanism of action of occlusive dressings in scarring. Wound Repair Regen. 2011 Sep;19 Suppl 1(0 1):s16-21. doi: 10.1111/j.1524-475X.2011.00709.x. PMID 21793961
- [Background] Steinstraesser L, Flak E, Witte B, Ring A, Tilkorn D, Hauser J, Langer S, Steinau HU, Al-Benna S. Pressure garment therapy alone and in combination with silicone for the prevention of hypertrophic scarring: randomized controlled trial with intraindividual comparison. Plast Reconstr Surg. 2011 Oct;128(4):306e-313e. doi: 10.1097/PRS.0b013e3182268c69. PMID 21921743
- [Background] Bloemen MC, van der Veer WM, Ulrich MM, van Zuijlen PP, Niessen FB, Middelkoop E. Prevention and curative management of hypertrophic scar formation. Burns. 2009 Jun;35(4):463-75. doi: 10.1016/j.burns.2008.07.016. Epub 2008 Oct 31. PMID 18951704

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total Started = 14. Each participant in the study received both treatment options (2 wounds per patient - one got treated with KeraStat Gel, one got treated with Silver Sulfadiazine).
Units Other Than Participants: Wounds
Groups:
- All Participants: Each enrolled subject will have two eligible burns. One burn will be randomly assigned to the KeraStat Gel arm of the study, and the other intrabody burn will be assigned to the SSD arm of the study. The KeraStat Gel area of injury will be dressed with KeraStat Gel and covered by a secondary dressing. The SSD area of injury will be dressed with SSD and covered by a secondary dressing. Subjects will be instructed to change the dressings per instructions for use.
Period: Overall Study
Arm/Group | All Participants
Started (Each subject received KeraStat Gel as well as Silver Sulfadiazine. Total subjects enrolled was 14, not 28.) | 14; 28 Wounds
KeraStat Gel-treated: (One (of two) wounds present on enrolled participants was treated with KeraStat Gel.) | 14; 14 Wounds
Silver Sulfadiazine-treated: (One (of two) wounds present on enrolled participants was treated with SSD.) | 14; 14 Wounds
Completed (Each subject received KeraStat Gel and Silver Sulfadiazine. Total number of subjects that completed the study was 3, not 6.) | 3; 6 Wounds
Not Completed | 11; 22 Wounds
Not completed — Withdrawal by Subject | 3
Not completed — Lost to Follow-up | 6
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Each enrolled subject will have at least one eligible burn randomized to the KeraStat Gel arm and SSD arm. The KeraStat Gel area of injury will be dressed with KeraStat Gel and covered by a secondary dressing. The SSD area of injury will be dressed with SSD and covered by a secondary dressing. Subjects will be instructed to change the dressings per instructions for use.
Arm/Group | All Participants
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 13
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.07 (16.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Improved Cosmesis
Description: The degree of cosmetic improvement of the healed wound will be assessed by Patient and Observer Scar Assessment Scale (POSAS) at one year. This scale consists of two parts: a Patient Scale and an Observer Scale. Both scales contain six items that are scored numerically on a 10-point range, where a '10' indicates the 'worst possible' [e.g. itching or pigmentation] and a '1' indicates normal skin. The Patient Scale is summed to make a 'Total Patient Score" ranging from 6 - 60. The Observer Scale is summed to make up a 'Total Observer Score' ranging from 6 - 60. The Total Patient Score and Total Observer Score can be summed into a Total POSAS Score ranging from 12 to 120.
Time Frame: One year post burn
Population: Each subject received both KeraStat Gel and Silver Sulfadiazine.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KeraStat Gel | Silver Sulfadiazine
Number analyzed (Participants) | 14 | 14
score on a scale
  POSAS - Observer (3 Month) | 12 (5.86) | 12.125 (5.62)
  POSAS - Observer (6 Month) | 10 (3.24) | 10 (2.92)
  POSAS - Observer (12 Month) | 7.67 (2.89) | 6 (4.36)
  POSAS - Patient (3 Month) | 4.125 (2.85) | 4.875 (2.95)
  POSAS - Patient (6 Month) | 5.4 (4.34) | 5.2 (4.09)
  POSAS - Patient (12 Month) | 6 (4.36) | 4.67 (3.51)

2. Secondary Outcome: Pain During Dressing Change
Description: Subject will complete Visual Analog Pain Scale (VAS) before and after in-clinic dressing changes. The Visual Analog Scale is presented as a 10 cm horizontal line ranging from 'No Pain' (0 cm) to 'Worst Pain Imaginable' (10 cm). The patient will mark the line to represent his or her level of pain before and after dressing changes.
Time Frame: Period during first month when dressing changes are required (Day 0, Day 7, Day 14, Day 21, Day 28).
Population: Each participant received KeraStat Gel and Silver Sulfadiazine.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 14
score on a scale
  Day 0 - Pain Score Immediately Prior to Dressing Change - KeraStat Gel | 3.14 (3.74)
  Day 0 - Pain Score Immediately Prior to Dressing Change - SSD | 2.86 (3.39)
  Day 0 - Pain Score During Dressing Change - KeraStat Gel | 4.14 (3.51)
  Day 0 - Pain Score During Dressing Change - SSD | 4.00 (3.46)
  Day 0 - Pain Score Immediately Following Dressing Change - KeraStat Gel | 4.14 (3.68)
  Day 0 - Pain Score Immediately Following Dressing Change - SSD | 3.64 (3.32)
  Day 0 - Pain Score 15 Minutes After Dressing Change - KeraStat Gel | 4.07 (3.38)
  Day 0 - Pain Score 15 Minutes After Dressing Change - SSD | 3.42 (2.93)
  Day 7 - Pain Score Immediately Prior to Dressing Change - KeraStat Gel: number analyzed (Participants) | 7
  Day 7 - Pain Score Immediately Prior to Dressing Change - KeraStat Gel | 2.57 (3.55)
  Day 7 - Pain Score Immediately Prior to Dressing Change - SSD: number analyzed (Participants) | 7
  Day 7 - Pain Score Immediately Prior to Dressing Change - SSD | 3.00 (3.70)
  Day 7 - Pain Score During Dressing Change - KeraStat Gel: number analyzed (Participants) | 7
  Day 7 - Pain Score During Dressing Change - KeraStat Gel | 3.86 (4.34)
  Day 7 - Pain Score During Dressing Change - SSD: number analyzed (Participants) | 7
  Day 7 - Pain Score During Dressing Change - SSD | 4.00 (4.32)
  Day 7 - Pain Score Immediately Following Dressing Change - KeraStat Gel: number analyzed (Participants) | 7
  Day 7 - Pain Score Immediately Following Dressing Change - KeraStat Gel | 3.29 (3.73)
  Day 7 - Pain Score Immediately Following Dressing Change - SSD: number analyzed (Participants) | 7
  Day 7 - Pain Score Immediately Following Dressing Change - SSD | 3.57 (3.95)
  Day 7 - Pain Score 15 Minutes After Dressing Change - KeraStat Gel: number analyzed (Participants) | 7
  Day 7 - Pain Score 15 Minutes After Dressing Change - KeraStat Gel | 2.71 (3.09)
  Day 7 - Pain Score 15 Minutes After Dressing Change - SSD: number analyzed (Participants) | 7
  Day 7 - Pain Score 15 Minutes After Dressing Change - SSD | 3.00 (3.37)
  Day 14 - Pain Score Immediately Prior to Dressing Change - KeraStat Gel: number analyzed (Participants) | 5
  Day 14 - Pain Score Immediately Prior to Dressing Change - KeraStat Gel | 1.80 (1.48)
  Day 14 - Pain Score Immediately Prior to Dressing Change - SSD: number analyzed (Participants) | 5
  Day 14 - Pain Score Immediately Prior to Dressing Change - SSD | 1.20 (1.10)
  Day 14 - Pain Score During Dressing Change - KeraStat Gel: number analyzed (Participants) | 5
  Day 14 - Pain Score During Dressing Change - KeraStat Gel | 2.00 (1.58)
  Day 14 - Pain Score During Dressing Change - SSD: number analyzed (Participants) | 5
  Day 14 - Pain Score During Dressing Change - SSD | 1.40 (1.34)
  Day 14 - Pain Score Immediately Following Dressing Change - KeraStat Gel: number analyzed (Participants) | 5
  Day 14 - Pain Score Immediately Following Dressing Change - KeraStat Gel | 1.90 (1.88)
  Day 14 - Pain Score Immediately Following Dressing Change - SSD: number analyzed (Participants) | 5
  Day 14 - Pain Score Immediately Following Dressing Change - SSD | 1.50 (1.50)
  Day 14 - Pain Score 15 Minutes After Dressing Change - KeraStat Gel: number analyzed (Participants) | 5
  Day 14 - Pain Score 15 Minutes After Dressing Change - KeraStat Gel | 1.70 (1.64)
  Day 14 - Pain Score 15 Minutes After Dressing Change - SSD: number analyzed (Participants) | 5
  Day 14 - Pain Score 15 Minutes After Dressing Change - SSD | 1.30 (1.48)
  Day 21 - Pain Score Immediately Prior to Dressing Change - KeraStat Gel: number analyzed (Participants) | 3
  Day 21 - Pain Score Immediately Prior to Dressing Change - KeraStat Gel | 1.00 (1.00)
  Day 21 - Pain Score Immediately Prior to Dressing Change - SSD: number analyzed (Participants) | 3
  Day 21 - Pain Score Immediately Prior to Dressing Change - SSD | 0.33 (0.58)
  Day 21 - Pain Score During Dressing Change - KeraStat Gel: number analyzed (Participants) | 3
  Day 21 - Pain Score During Dressing Change - KeraStat Gel | 1.00 (1.00)
  Day 21 - Pain Score During Dressing Change - SSD: number analyzed (Participants) | 3
  Day 21 - Pain Score During Dressing Change - SSD | 0.33 (0.58)
  Day 21 - Pain Score Immediately After Dressing Change - KeraStat Gel: number analyzed (Participants) | 3
  Day 21 - Pain Score Immediately After Dressing Change - KeraStat Gel | 1.00 (1.00)
  Day 21 - Pain Score Immediately After Dressing Change - SSD: number analyzed (Participants) | 3
  Day 21 - Pain Score Immediately After Dressing Change - SSD | 0.33 (0.58)
  Day 21 - Pain Score 15 Minutes After Dressing Change - KeraStat Gel: number analyzed (Participants) | 3
  Day 21 - Pain Score 15 Minutes After Dressing Change - KeraStat Gel | 1.00 (1.00)
  Day 21 - Pain Score 15 Minutes After Dressing Change - SSD: number analyzed (Participants) | 3
  Day 21 - Pain Score 15 Minutes After Dressing Change - SSD | 0.33 (0.58)
  Day 28 - Pain Score Immediately Prior to Dressing Change - KeraStat Gel: number analyzed (Participants) | 1
  Day 28 - Pain Score Immediately Prior to Dressing Change - KeraStat Gel | 1.00 (NA) — Insufficient participants to generate standard deviation.
  Day 28 - Pain Score Immediately Prior to Dressing Change - SSD: number analyzed (Participants) | 1
  Day 28 - Pain Score Immediately Prior to Dressing Change - SSD | 1.00 (NA) — Insufficient participants to generate standard deviation.
  Day 28 - Pain Score During Dressing Change - KeraStat Gel: number analyzed (Participants) | 1
  Day 28 - Pain Score During Dressing Change - KeraStat Gel | 1.00 (NA) — Insufficient participants to generate standard deviation.
  Day 28 - Pain Score During Dressing Change - SSD: number analyzed (Participants) | 1
  Day 28 - Pain Score During Dressing Change - SSD | 1.00 (NA) — Insufficient participants to generate standard deviation.
  Day 28 - Pain Score Immediately Following Dressing Change - KeraStat Gel: number analyzed (Participants) | 1
  Day 28 - Pain Score Immediately Following Dressing Change - KeraStat Gel | 1.00 (NA) — Insufficient participants to generate standard deviation.
  Day 28 - Pain Score Immediately Following Dressing Change - SSD: number analyzed (Participants) | 1
  Day 28 - Pain Score Immediately Following Dressing Change - SSD | 1.00 (NA) — Insufficient participants to generate standard deviation.
  Day 28 - Pain Score 15 Minutes After Dressing Change - KeraStat Gel: number analyzed (Participants) | 1
  Day 28 - Pain Score 15 Minutes After Dressing Change - KeraStat Gel | 1.00 (NA) — Insufficient participants to generate standard deviation.
  Day 28 - Pain Score 15 Minutes After Dressing Change - SSD: number analyzed (Participants) | 1
  Day 28 - Pain Score 15 Minutes After Dressing Change - SSD | 1.00 (NA) — Insufficient participants to generate standard deviation.

ADVERSE EVENTS:
Time Frame: Through study completion, up to 1 year
Groups:
- KeraStat Gel-treated Wound; Silver Sulfadiazine-treated Wound: Each enrolled subject will have 2 wounds. One wound will be randomized to the KeraStat Gel arm and the other will be assigned the Silver Sulfadiazine arm. The KeraStat Gel area of injury will be dressed with KeraStat Gel and covered by a secondary dressing. The SSD area of injury will be dressed with SSD and covered by a secondary dressing. Subjects will be instructed to change the dressings per instructions for use.
Arm/Group | KeraStat Gel-treated Wound | Silver Sulfadiazine-treated Wound
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-05): https://cdn.clinicaltrials.gov/large-docs/95/NCT03564795/Prot_SAP_001.pdf